CLINICAL TRIAL: NCT00537056
Title: Evaluating Sunitinib Therapy in Renal Cell Carcinoma Using F-18 FDG PET/CT and DCE MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Andrew Quon, Associate Professor of Radiology (Nuclear Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-08558; 97807 (Other: Stanford University Alternate IRB Approval Number); RENAL0013 (Other: OnCore)
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Kidney Neoplasms; Carcinoma, Renal Cell; Kidney (Renal Cell) Cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; Gadolinium DTPA; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F-18 FDG PET/CT and DCE MRI (Experimental): FDG PET CT F-18 Fluoro-deoxi-glucose: 15 mCi iv Gadolinium-DTPA: 0.1 mmol/kg Sunitinib: 50 mg/day po
  Interventions: Procedure: FDG PET CT; Procedure: DCE MRI; Drug: F-18 Fluoro-deoxi-glucose; Drug: Gadolinium-DTPA; Drug: Sunitinib

INTERVENTIONS:
Procedure: FDG PET CT — nuclear medicine imaging technique which produces a three-dimensional image or picture of functional processes in the body
  Other Names: Positron emission tomography (PET)
Procedure: DCE MRI — DCE MRI will be acquired using rapid intravenous bolus of gadolinium-DTPA (0.1 mmol/kg).
  Other Names: Magnetic Resonance Imaging
Drug: F-18 Fluoro-deoxi-glucose — 15 mCi iv
  Other Names: fluorodeoxyglucose (18F); Fludeoxyglucose (18F); 18F-FDG; FDG
Drug: Gadolinium-DTPA — 0.1 mmol/kg iv
  Other Names: Gadopentetic acid; gadopentetate dimeglumine; Gd-DTPA; Berlex
Drug: Sunitinib — 50 mg/day po
  Other Names: Sutent; SU11248

SUMMARY:
To learn whether Flourine-18 Fluoro-deoxi-glucose positron emission tomography / computed tomography (F-18 FDG PET/CT) and dynamic contrast enhanced magnetic resonance imaging (DCE MRI) are better predictors of response to therapy than the current standard of care (CT or MRI).

DETAILED DESCRIPTION:
This is a single arm prospective trial in patients with newly-diagnosed advanced renal cell cancer (RCC) who were scheduled for sunitinib therapy and utilized an extensive panel of quantitative metrics on baseline and interim FDG PET/CT to evaluate the predictive utility of each of these measurements.

The objectives were to evaluate the FDG PET/CT measurement parameters for prediction of prognosis after sunitinib therapy in patients with RCC using histopathologic (post-therapy nephrectomy) or clinical follow-up for validation.

ELIGIBILITY:
Inclusion Criteria:- Measurable disease by RECIST criteria

* Pathologic diagnosis of renal cell cancer
* Advanced (stage IV) renal cell cancer
* Karnofsky performance status of (KPS>70)
* Consent to participate in the clinical trial Exclusion Criteria:- Patients who cannot complete a PET/CT scan.
* Pregnant women.
* Healthy volunteers.
* Patients participating in other research protocols will be excluded from this study.
* Metallic implants (prosthesis, ICD, pacemakers), since these are contraindications for MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-10; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Andrew Quon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified (anonymized) patient data is routinely provided upon request. Protecting patient privacy and confidentiality is the utmost consideration when sharing individual patient data. In all cases of data sharing, patient data is always anonymized to protect privacy. All potential identifiers (name, hospital ID, address,etc) are removed.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventeen previously untreated adult patients with advanced stage IV renal cell carcinoma (RCC) were prospectively recruited to Stanford Hospital and Clinics for a baseline PET/CT scan followed by a 12-month follow-up PET/CT scan post sunitinib therapy.
Groups:
- F-18 FDG PET/CT and DCE MRI: 15 mCi iv F-18 FDG PET/CT scan and DCE MRI using Gadolinium-DTPA: 0.1 mmol/kg iv followed by Sunitinib therapy at 50 mg/day.
Period: Baseline PET/CT
Arm/Group | F-18 FDG PET/CT and DCE MRI
Started | 17
Completed | 17
Not Completed | 0
Period: Interim PET/CT
Arm/Group | F-18 FDG PET/CT and DCE MRI
Started | 17
Completed | 12
Not Completed | 5
Not completed — scheduling conflicts and/or exposure | 5
Period: 12-month Follow-up
Arm/Group | F-18 FDG PET/CT and DCE MRI
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants] — Stanford Hospital and Clinics
  participants
    United States | 17

OUTCOME MEASURES:

1. Primary Outcome: F-18 FDG Tumor Uptake (SUV Max)
Description: The maximum standardized uptake value (SUVmax) is a measurement of tumor metabolism as determined by the PET scan before and after 12-weeks of sunitinib therapy. Decreased SUVmax correlates to a reduction of tumor metabolism. Increased SUVmax correlates to an increase in tumor metabolism.
  Reduction or increased SUVmax will be determined as the change from baseline in uptake of F18 FDG.
  Results were based on the European Organization for Research and Treatment of Cancer (EORTC) for predicting progression free survival. EORTC criteria is a ± 25% change of SUVmax for assessment of progressive disease, stable disease and partial response.
Time Frame: 12 weeks minus baseline
Population: All patients underwent baseline F-18 FDG PET scan. Mean SUVmax at baseline is reported (row 1). 6 participants achieved progression-free survival after post-sunitinib therapy, and their SUVmax values were averaged (row 2). 11 participants had progression or recurrence/relapse of disease and their SUVmax values were averaged (row 3).
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- F-18 FDG PET/CT and DCE MRI: 15 mCi iv F-18 FDG PET/CT scan
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
SUVmax
  Baseline SUVmax | 9.8 (5.7)
  Mean SUVmax, progression-free survival: number analyzed (Participants) | 6
  Mean SUVmax, progression-free survival | -18.9 (15.1)
  SUVmax, progression/relapse: number analyzed (Participants) | 11
  SUVmax, progression/relapse | 34.0 (39.7)

2. Secondary Outcome: Histopathology
Description: Histopathologic findings were correlated to the pre-treatment 18F-fluorodeoxyglucose positron emission tomography (F-18 FDG PET/CT) scan. Outcome is reported as the number of participants for whom both histopathology and F-18 FDG PET/CT indicated that active cancers was present.
Time Frame: 1 day
Population: Patients with renal cell carcinoma
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | 17

3. Secondary Outcome: Initial Comprehensive Metabolic Panel
Description: A comprehensive metabolic panel is a blood test that measures sugar (glucose) level, electrolyte and fluid balance, kidney function, and liver function. It was performed prior to the administration of gadolinium contrast. For patients with normal renal function, approximately 90% of gadolinium contrast is excreted through the urinary system. These patients have known renal cell carcinoma, so it was important to perform a metabolic function panel prior to gadolinium injection, specifically to determine kidney function. Reported as the number of patients for whom the initial comprehensive metabolic panel was within institutional standards.
Time Frame: Prior to baseline DCE MRI
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | 17

4. Secondary Outcome: Adverse Events
Description: Adverse events were monitored for on F-18 FDG PET/CT and DCE MRI imaging days: baseline (n=17); interim (n=12); and post-sunitinib therapy (n=17). Reported as the overall number of adverse events experienced.
Time Frame: up to 12 months
Measure: Number; unit: adverse events
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
adverse events | 0

5. Secondary Outcome: Tumor Necrosis
Description: The degree of tumor necrosis was measured using values obtained from dynamic contrast enhanced magnetic resonance imaging (DCE MRI) pre- and post-sunitinib therapy. Gadolinium contrast material given intravenously during the DCE MRI scan is used to improve visualization of blood vessels, tumors, and/or organs.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | NA — The DCE MRI image was obtained but image quality was poor and the degree of tumor necrosis could not be determined.

6. Secondary Outcome: Tumor Size by Computed Tomography (CT) Scan
Description: Tumor size was measured based on computed tomography (CT) pre- and post-sunitinib therapy. CT was performed immediately prior to the PET scan and is used to determine both the PET scan imaging area and PET image attenuation correction (AC). F-18 FDG PET provides the metabolic and physiologic data while CT provides the anatomical data.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- F-18 FDG PET/CT and DCE MRI: 15 mCi iv F-18 FDG PET/CT scan followed by Sunitinib therapy at 50 mg/day.
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | NA — The CT scan performed immediately prior to the PET scan was of poor (non-diagnostic) quality and did not provide usable size measurement data.

7. Secondary Outcome: Tumor Size by DCE Magnetic Resonance Imaging (MRI) Scan
Description: Tumor size was measured using values obtained from DCE MRI pre- and post-sunitinib therapy. Gadolinium contrast material given intravenously during the DCE MRI scan is used to improve visualization of blood vessels, tumors, and/or organs.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | NA — The DCE MRI image was obtained but image quality was poor and provided no useful data from which to determine tumor size.

8. Secondary Outcome: DCE MRI AUC Peak Flow
Description: Area under the curve (AUC) was measured using receiver operating characteristic (ROC) curve analysis. ROC curve analysis measures sensitivity (true-positives, correctly diagnosed positive pathologies) against specificity (true-negatives, correctly diagnosed negative pathologies or free of disease) of the DCE MRI scan. An area of 1.0 under the curve would equal a perfect test (with 100% sensitivity; 100% specificity) while an area of 0.5 would equal a useless test (50% sensitivity; 50% specificity).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | NA — The DCE MRI image was obtained but image quality was poor and provided no useful data to determine AUC.

9. Secondary Outcome: Initial Tumor Size
Description: Initial tumor size was measured using values obtained from computed tomography (CT) pre-sunitinib therapy. CT is performed immediately prior to the PET scan and is used to determine both the PET scan imaging area and PET image attenuation correction (AC). F-18 FDG PET provides the metabolic and physiologic data while CT provides the anatomical data.
Time Frame: pre-sunitinib therapy
Measure: Count of Participants; unit: Participants
Arm/Group | F-18 FDG PET/CT and DCE MRI
Number analyzed (Participants) | 17
Participants | NA — The CT scan performed immediately prior to the PET scan was of poor image quality (non-diagnostic) and did not provide usable measurement data.

ADVERSE EVENTS:
Time Frame: up to 12 months
Description: No adverse events were noted, and none are reported.
Arm/Group | F-18 FDG PET/CT and DCE MRI
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
The utility of the MRI- and CT-scans was significantly limited by low image quality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No